CLINICAL TRIAL: NCT01211665
Title: High-Dose Corticosteroids for Immune Reconstitution Inflammatory Syndrome in Patients Who Develop Progressive Multifocal Leukoencephalopathy on Natalizumab
Brief Title: Corticosteroids for Immune Reconstitution Inflammatory Syndrome (IRIS)
Acronym: IRIS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped prematurely due to lack of enrollment within a 1-5-year period.
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101JC404; 2010-020369-26 (EudraCT Number)
Record Dates: First submitted 2010-07-29; First posted 2010-09-29 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Immune Reconstitution Inflammatory Syndrome; Leukoencephalopathy, Progressive Multifocal
Keywords: IVMP; corticosteroids; IRIS; Progressive Multifocal Leukoencephalopathy; Immune reconstitution inflammatory syndrome; PML
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; Leukoencephalopathy, Progressive Multifocal | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisolone

ARMS (2):
- Pulsed IVMP (Experimental): Intravenous methylprednisolone (IVMP) 1 g/day administered the first 3 days of each weekly cycle, and repeated for 3 additional cycles (totaling 4 cycles). If necessary, 2 additional weekly cycles of 1 g IVMP daily for 3 days can be administered at the discretion of the investigator.
  Interventions: Drug: Methylprednisolone
- IVMP with oral prednisolone taper (Experimental): Intravenous methylprednisolone (IVMP) 1g/day for 6 days followed by an oral taper of prednisolone over 2 months (suggested dosages starting at 80 mg and tapering to 5 mg). If necessary, additional cycles of 1 g IVMP daily for 3 to 5 days can be administered at any time.
  Interventions: Drug: Methylprednisolone; Drug: Prednisolone

INTERVENTIONS:
Drug: Methylprednisolone — In intravenous form (for a daily dose of 1 g/day on treatment days).
  Other Names: Medrol; Solu-Medrol
Drug: Prednisolone — Oral prednisolone used as a taper, with suggested dosages starting at 80 mg and tapering to 5 mg.
  Other Names: Orapred; Prelone
  Arms: IVMP with oral prednisolone taper

SUMMARY:
The objectives of this study are to explore the effects of administering high-dose corticosteroids to participants who developed progressive multifocal leukoencephalopathy (PML) while on natalizumab as measured by time-course change in functional status based on Karnofsky Performance Status Index through 6 months following the completion of plasma exchange (PLEX; or equivalent), survival at 6 months following the completion of PLEX (or equivalent), and incidence and severity of adverse events (AEs) and serious adverse events (SAEs); to characterize the evolution of immune reconstitution inflammatory syndrome (IRIS) as measured by time course changes in Global Clinical Impression of Improvement (GCI-I), Symbol Digit Modalities Test (SDMT), brain magnetic resonance imaging (MRI), magnetoencephalography (MEG), chemokines, cytokines, C-reactive protein (CRP), John Cunningham virus (JCV) load and cell count in cerebrospinal fluid (CSF); and to characterize the time course elimination of serum natalizumab concentrations in the study population following the last PLEX (or equivalent) procedure.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have been receiving natalizumab for multiple sclerosis (MS) prior to the diagnosis or suspicion of Progressive multifocal leukoencephalopathy (PML).
* Subject must be willing to undergo or have completed plasma exchange (PLEX) prior to initiating study treatment.

Key Exclusion Criteria:

* History of severe allergic or anaphylactic reactions or known hypersensitivity to any drug including hypersensitivity to corticosteroids.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- Research Site, Hastings, Nebraska, United States
- Germany (2):
  - Research Site, Bochum
  - Research Site, Würzburg

RESULTS

PARTICIPANT FLOW:
Groups:
- IVMP With Oral Prednisolone Taper: Intravenous methylprednisolone (IVMP) 1g/day for 6 days followed by an oral taper over 2 months. If necessary, additional cycles of 1 g IVMP daily for 3 to 5 days can be administered at any time.
Period: Overall Study
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Started | 2 | 1
Completed | 0 | 1 (completed treatment with study drug)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time Course Change in Functional Status Based on Karnofsky Performance Status Index Through 6 Months Following Completion of Plasma Exchange (PLEX)
Description: The Karnofsky Performance Status Index (KPSI) is an assessment tool intended to assist clinicians and caretakers in gauging a patient's functional status and ability to carry out activities of daily living. A KPSI of 100=normal, no complaints, no evidence of disease; 90=able to carry on normal activity, minor signs or symptoms of disease; 80=normal activity with effort, some signs or symptoms of disease; 70=cares for self, unable to carry on normal activity or do active work; 60=requires occasional assistance but is able to care for most personal needs; 50=requires considerable assistance and frequent medical care; 40=disabled, requires special care and assistance; 30=severely disabled, hospitalization is indicated, although death is not imminent; 20=very sick, hospitalization is necessary, active support treatment is necessary; 10=moribund, fatal processes progressing rapidly; 0=dead.
Time Frame: Baseline up to 6 months
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants Who Survived at 6 Months Following Completion of Plasma Exchange (PLEX)
Description: Following the completion of rapid removal of natalizumab using PLEX or equivalent.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 2 | 1
participants | 1 | 1

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE=any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: from the first dose of study treatment through the end of the treatment period (6 months) + a 4-week post-treatment period
Measure: Number; unit: participants
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 2 | 1
participants
  AEs | 2 | 1
  SAEs | 2 | 1

4. Primary Outcome: Severity of AEs and SAEs
Description: AEs and SAEs were categorized as mild, moderate or severe according to the following criteria: Mild=barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptom(s) but may be given because of personality of participant. Moderate=of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptom(s) may be needed. Severe=symptoms cause severe discomfort; symptoms cause incapacity or significant impact on participant's daily life; severity may cause cessation of treatment with study treatment; treatment for symptom(s) may be given and/or participant hospitalized. Please see Outcome Measure 3 for AE and SAE definitions.
Time Frame: as for outcome 3
Measure: Number; unit: events
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 2 | 1
events
  Mild SAE | 1 | 1
  Moderate SAE | 1 | 1
  Severe SAE | 2 | 0
  Mild AE | 3 | 5
  Moderate AE | 3 | 1
  Severe AE | 0 | 0

5. Primary Outcome: Time Course Change in the Global Clinical Impression of Improvement (GCI-I) Scale
Description: The GCI-I scale is a 7-point scale that assesses how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention, and rates it as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Screening to 6 months following completion of PLEX (participants began treatment with intravenous methylprednisolone (IVMP) within 2 weeks after PLEX [or equivalent]).
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Time Course Change in Cerebral Dysfunction Using the Symbol Digit Modalities Test (SDMT)
Description: The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution.
Time Frame: Screening to 6 months following completion of PLEX (participants began treatment with IVMP within 2 weeks after PLEX [or equivalent]).
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Time Course Changes in Brain Magnetic Resonance Imaging (MRI)
Description: The brain MRI data collected included: progressive multifocal leukoencephalopathy (PML) lesion localization, T2 hyperintense lesion volume, and signs of cerebral edema.
Time Frame: as for outcome 6
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Time Course Change in Magnetoencephalography (MEG) Results
Description: MEG was used to map brain activity.
Time Frame: as for outcome 6
Population: This study was stopped prematurely due to lack of enrollment; no data on this endpoint was collected.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Time Course Change in Clinical Laboratory Values
Description: Clinical laboratory values included chemokines, cytokines, C-reactive protein (CRP), John Cunningham (JC) virus load, and cell count in cerebrospinal fluid.
Time Frame: as for outcome 6
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Time Course Elimination of Serum Natalizumab Concentration Following Plasma Exchange (PLEX) or Equivalent
Time Frame: Baseline up to 6 months
Population: This study was stopped prematurely due to lack of enrollment; this analysis was not performed.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the first dose of study treatment through the end of the treatment period (6 months) + a 4-week post-treatment period.
Arm/Group | Pulsed IVMP | IVMP With Oral Prednisolone Taper
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulsed IVMP (N=2) | IVMP With Oral Prednisolone Taper (N=1)
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune Reconstitution Syndrome (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulsed IVMP (N=2) | IVMP With Oral Prednisolone Taper (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.